CLINICAL TRIAL: NCT05310929
Title: Nitroglycerin Versus Labetalol in Acute Severe Pre-eclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R47/2019
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Severe Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Labetalol; Nitroglycerin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N ( nitroglycerine group ) (Experimental): Group N received nitroglycerin intravenous infusion in a concentration of 1 mg/ml, thus 1µg/Kg/min equals to 4.8 ml/hr for an 80 Kg patient. The infusion rate was titrated to stabilize systolic blood pressure (SBP) at 130-140 mmHg and diastolic blood pressure (DBP) at 80-90 mmHg (study end point) by adjusting the infusion rate as required either by maintaining the same infusion rate or by changing its infusion rate by 1 ml/hr up or down according to the clinical condition every 10 minutes.
  Interventions: Drug: Labetalol and Glyceril trinitrate
- Group L (labetalol group) (Experimental): . Group L received labetalol intravenous infusion in a concentration of 10 mg/ ml, thus 50 mg/ml equals to 5 ml/hr. The starting infusion rate of the antihypertensive medication was 5 ml/hr. The infusion rate was titrated to stabilize systolic blood pressure (SBP) at 130-140 mmHg and diastolic blood pressure (DBP) at 80-90 mmHg (study end point) by adjusting the infusion rate as required either by maintaining the same infusion rate or by changing its infusion rate by 1 ml/hr up or down according to the clinical condition every 10 minutes.
  Interventions: Drug: Labetalol and Glyceril trinitrate

INTERVENTIONS:
Drug: Labetalol and Glyceril trinitrate — for control of blood pressure
  Other Names: Trandate and nitroglycerin

SUMMARY:
Two hundred patients with severe PE were admitted prepartum to the ICU to stabilize blood pressure. They were randomly assigned to one of two groups (100 in each group): Group N received nitroglycerine intravenous infusion in a concentration of 1 mg/ml, thus 1µg/Kg/min equals to 4.8 ml/hr for an 80 Kg patient. Group L received labetalol intravenous infusion in a concentration of 10 mg/ ml, thus 50 mg/ml equals to 5 ml/hr. The starting infusion rate of the antihypertensive medication was 5 ml/hr. The infusion rate was titrated to stabilize systolic blood pressure (SBP) at 130-140 mmHg and diastolic blood pressure (DBP) at 80-90 mmHg (study end point) by adjusting the infusion rate as required either by maintaining the same infusion rate or by changing its infusion rate by 1 ml/hr up or down according to the clinical condition every 10 minutes. On any abrupt reduction in blood pressure below 120 mmHg for SBP or 80 mmHg for DBP, the infusion was immediately discontinued, and a bolus of 150 ml lactate ringer was given.

DETAILED DESCRIPTION:
Patients and Methods The study was conducted in the intensive care unit (ICU) of the Obstetrics and Gynaecology Hospital of Ain-Shams University as a randomized, double-blind, and placebo-controlled study on patients diagnosed with severe PE from July 2016 to June 2018. The study was approved by Ethical Research Committee at Ain Shams University (ethical number FMASU R 47/2019) and all participants provided written informed consent.

Woman eligible for this study were aged between 18-40 years old at greater than 34 weeks of gestation having severe PE without severe features (without imminence of eclampsia or clinical manifestations of target organ damage, as per the ACOG criteria) (7). Severe PE was diagnosed by severe hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg, repeated measurement should be taken for confirmation no more than 15 minutes later), presence of clinically significant proteinuria (0.3 grams or more of protein in 24-hour urine collection, or urinary protein/creatinine ratio of 30 or more)[8].

Exclusion criteria were patients with chronic hypertension, imminence of eclampsia, target organ damage, active asthma and congestive heart failure. Patients with any known allergy to one of the study drugs are also excluded.

Two hundred patients with severe PE were admitted prepartum to the ICU to stabilize blood pressure. They were randomly assigned to one of two groups (100 in each group): Group N received nitroglycerine intravenous infusion in a concentration of 1 mg/ml, thus 1µg/Kg/min equals to 4.8 ml/hr for an 80 Kg patient. Group L received labetalol intravenous infusion in a concentration of 10 mg/ ml, thus 50 mg/ml equals to 5 ml/hr. The starting infusion rate of the antihypertensive medication was 5 ml/hr. The infusion rate was titrated to stabilize systolic blood pressure (SBP) at 130-140 mmHg and diastolic blood pressure (DBP) at 80-90 mmHg (study end point) by adjusting the infusion rate as required either by maintaining the same infusion rate or by changing its infusion rate by 1 ml/hr up or down according to the clinical condition every 10 minutes. On any abrupt reduction in blood pressure below 120 mmHg for SBP or 80 mmHg for DBP, the infusion was immediately discontinued, and a bolus of 150 ml lactate ringer was given.

Randomization was attained by using orderly numbered, opaque sealed envelopes containing computer-generated random allocations.

Patients received full intensive care treatment for PE according to the standard protocol of the obstetric ICU of Ain-Shams University. All treatments were provided by physicians who were not involved in the study including infusion of lactated Ringer solution at a starting rate of 75 ml/hr and then adjusted according to the fluid balance, magnesium sulfate (4 gm IV loading dose over a period of 10 minutes and 1 gm/hr IV infusion until 24 hours after delivery as seizure prophylaxis, its dose was adjusted according to renal function) in addition to antihypertensive medications according to the assigned group. The study solution was stopped if maternal pulse reached less than 60 bpm or increased more than 110 bpm.

Vital signs were monitored at admission and until patients were discharged from the ICU using ECG, pulse oximetry, continuous invasive arterial blood pressure monitoring through radial artery, and an indwelling catheter for urine output assessment.

Assessment of fetal well-being was done before starting of the study in the form of cardiotocography (CTG), modified biophysical profile, doppler US on umbilical artery, and growth scan. In addition, continuous fetal heart rate monitoring was done by CTG during the study time.

Severe persistent hypertension was considered when SBP was greater than 160 mmHg or DBP was greater than 110 mmHg after the administration of maximum dose of allocated drug treatment; 20 ml/hr. Hence, patient was shifted to sodium nitroprusside infusion after 2 hours of starting treatment with assigned drugs.

After stabilization of the patient and once the target BP was achieved, induction of labor was started using 3 mg prostaglandin E2 (PGE2) vaginal tablet. It was to be repeated after 6 hours if needed. In case oxytocin was to be used, it was administered at least 6 hours apart from PGE2 last dose.

If the patient was not eligible for induction of labor as in case of previous cesarean delivery (CS), transverse lie of the fetus and other standard obstetrical indications, CS was done at once. CS was also performed in case of failed induction of labor (no uterine contractions nor cervical changes after 6mg of PGE2), fetal compromise, arrest of progress of labor, arrest of cervical dilatation, arrest of fetal descent, and in case of moderate or severe accidental hemorrhage.

The following data were recorded and included demographic characteristics, the time taken to control blood pressure (time from starting infusion till reaching study end point), and number of sudden attacks of hypotension (BP values below the desired level). In addition, side effects of drugs such as tachycardia (HR>100 bpm), bradycardia HR<60 bpm) headache, nausea/vomiting, hypotension, flushing, dizziness were recorded. The mode of delivery either vaginal or caesarean section was also recorded. Fetal outcome regarding stillbirths (death in utero at or after 20 weeks' gestation) and suspected fetal compromise by abnormal CTG (continuous or progressive fetal bradycardia <100 bpm, reduced fetal heart rate variability (<5 bpm) that last more than 90 minutes, atypical variable decelerations with over 50% of contractions, late decelerations for >30 minutes, single prolonged decelerations for more than 3 minutes, or sinusoidal pattern more than 10 minutes). 1 min Apgar score less than 7- and 5-minutes Apgar score less than 7 were also recorded.

ELIGIBILITY:
Inclusion Criteria:Woman eligible for this study were aged between 18-40 years old at greater than 34 weeks of gestation having severe PE without severe features (without imminence of eclampsia or clinical manifestations of target organ damage, as per the ACOG criteria) (7). Severe PE was diagnosed by severe hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg, repeated measurement should be taken for confirmation no more than 15 minutes later), presence of clinically significant proteinuria (0.3 grams or more of protein in 24-hour urine collection, or urinary protein/creatinine ratio of 30 or more) -

Exclusion Criteria:patients with chronic hypertension, imminence of eclampsia, target organ damage, active asthma and congestive heart failure. Patients with any known allergy to one of the study drugs are also excluded.

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females having pre eclampsia
Enrollment: 200 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
time required to control blood pressure by the assigned group | within 2 hours from start of therapy
  The infusion rate was titrated to stabilize systolic blood pressure (SBP) at 130-140 mmHg and diastolic blood pressure (DBP) at 80-90 mmHg (study end point)

CONTACTS AND LOCATIONS:
Overall Officials: Fathy Tash, MD, Study Chair — Ain Shams University
Locations (1):
- AinShams university hospitals, Cairo, Egypt